CLINICAL TRIAL: NCT04497740
Title: Retrospective Evaluation of Follow-up Results of Newborns Who Underwent Tracheostomy
Brief Title: Follow-up Results of Newborns With Tracheostomy
Acronym: FRONWT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, H. Tolga Çelik, associate professor, Hacettepe University
Other Study IDs: GO20529
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Premature; Tracheostomy Complication; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The chances of survival in premature babies, especially in babies born under 28 weeks, have increased in recent years, and comorbidities also increase. Bronchopulmonary dysplasia (BPD), one of the premature problems, is one of them. After a while, babies with heavy BPD are discharged with the support of a home-type mechanical ventilator by opening a tracheostomy. Tracheostomy procedure is performed by specialist doctors of otolaryngology under general anesthesia in the operating room conditions in newborns. Complications of this procedure such as bleeding, skin necrosis, decanulation, trachea laceration and infection in the early period can be seen. In the long term, in addition to complications such as formation of tracheal granulation tissue, ulceration, laceration due to the procedure, babies with tracheostomy may develop nutrition and speech problems and neurodevelopmental problems.

In the literature, there is no comprehensive clinical follow-up study involving early and late clinical results related to newborns undergoing tracheostomy. In this study, early and late follow-up results (indications, anthropometric measurements, mechanical ventilation and oxygen deposition times, complications, tracheostomy closure times, tracheostomy closure times, neurodevelopmental patients in the Neonatal Intensive Care Unit of Hacettepe University Ihsan Dogramaci Children's Hospital. results, accompanying other comorbidities, etc.).

DETAILED DESCRIPTION:
With the advances in science and technology in recent years, the rate of survival of high-risk newborns has increased in neonatal intensive care units. Some of these babies are left in the neonatal intensive care unit for a long time, and because of the need for respiratory support, tracheostomy is opened and discharged with home mechanical ventilator devices.

Especially babies with severe BPD cannot be extubated and they may be exposed to trauma of long-term intubation. Subglottic stenosis is the most common result of this trauma. Some of the babies with severe BPD are discharged by the otolaryngology specialist doctor before discharge, to prevent both long-term intubation complications, airway obstruction or tracheal stenosis and adaptation to the home mechanical ventilator.

In addition to babies with BPD, tracheostomy is opened to babies in the early period due to various developmental tracheal anomalies in our unit. Some of these are congenital tracheal stenosis, congenital laryngeal atresia, laryngeal web.

In the following process, the growth of the baby, the development of the lungs and auxiliary respiratory muscles and the need for mechanical ventilator support are eliminated and the patient can wean from the ventilator support. In addition, the tracheostomy procedure secures the patient's airway and allows it to be fed easily by mouth and the comfort of the patient.

When the tracheostomy requirement of the patient disappears (mechanical ventilator, when oxygen is not needed), tracheostomy closure can be performed to ensure the patient has normal larynx functions (sounding, speech, airway protection reflexes).

In the literature, there is no comprehensive clinical follow-up study involving early and late clinical results related to newborns undergoing tracheostomy. In this study, early and late follow-up results (indications, anthropometric measurements, mechanical ventilation and oxygen deposition times, complications, tracheostomy closure times, tracheostomy closure times, neurodevelopmental patients in the Neonatal Intensive Care Unit of Hacettepe University Ihsan Dogramaci Children's Hospital results, accompanying other comorbidities, etc.). This study is planned as a retrospective study. Participants planned to determine the results of the study whether these babies should be careful in the follow-up and to take precautions in order to lead a better and healthier life, and what participants can do in order to provide these babies and their families with better health care support.

ELIGIBILITY:
Inclusion Criteria:

* These are the babies who stayed in Hacettepe University Ihsan Dogramaci Children's Hospital Neonatal Intensive Care Unit between 01.01.2005-31.12.2019, underwent tracheostomy procedure and followed up at risky neonatal outpatient clinic.

Exclusion Criteria:

* Newborns whose file and follow-up information required for the study are not available

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: These are the babies who stayed in Hacettepe University Ihsan Dogramaci Children's Hospital Neonatal Intensive Care Unit between 01.01.2005-31.12.2019, underwent tracheostomy procedure and followed up at risky neonatal outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-08-10 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
follow up after tracheostomy | 15 years
  Follow-up of patients who have been in our NICU for the last fifteen years and discharged with tracheostomy.

SECONDARY OUTCOMES:
evaluation of tracheostomy opening indications | 15 years
  indications of tracheostomy in the last fifteen years in our unit

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tandircioglu UA, Dogan O, Gunaydin RO, Yigit S, Celik HT. Outcomes of newborns with tracheostomy: single center experience. Turk J Pediatr. 2023;65(4):555-561. doi: 10.24953/turkjped.2023.185. PMID 37661670
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30396419/

DOCUMENTS (1):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT04497740/Prot_000.pdf